CLINICAL TRIAL: NCT00867581
Title: To Observe Delayed Neuronal Death of Hippocampus After Middle Cerebral Artery Infarction Through Magnetic Resonance Imaging(MRI) Volume Measurement and Magnetic Resonance Spectroscopy(MRS) Study of Hippocampus
Brief Title: Magnetic Resonance Imaging (MRI) Study of the Hippocampus After Infarction in the Territory of the Middle Cerebral Artery
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Huazhong University of Science and Technology (Other)
Responsible Party: Wei Wang, Department of Neurology of Tongji Hospital, Huazhong University of Sci. and Tec
Other Study IDs: 30725019-2
Record Dates: First submitted 2009-03-23; First posted 2009-03-24 (Estimated); Last update posted 2009-03-24 (Estimated); Status verified 2009-03

CONDITIONS: Ischemic Stroke
Keywords: middle cerebral artery; infarction; chronic stage; hippocampal volume; MRI; MRS; neuropsychologic assessment
MeSH Terms: conditions — Ischemic Stroke; Infarction

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Cross-Sectional
Oversight: Data Monitoring Committee: Yes

GROUPS / COHORTS (2):
- 1: chronic-stage patients after infarction in the territory of unilateral middle cerebral artery
- 2: age, sex and risk factor matched volunteers without ischemic stroke

SUMMARY:
The purpose of this study is to observe delayed neuronal death of hippocampus after middle cerebral artery infarction in human beings.

DETAILED DESCRIPTION:
40 patients with middle cerebral artery infarction and 40 healthy volunteers will be observed. All of them will receive MRI scan and the assessment of the neuropsychological function (MMSE, AVLT, HAMD) intending to observe delayed neuronal death of hippocampus after middle cerebral artery infarction in human beings.

ELIGIBILITY:
Inclusion Criteria:

* Clinical diagnosis of middle cerebral artery infarction
* At least six months from the stroke
* Must be able to measure his(her) neuropsychologic function (by MMSE, AVLT)

Exclusion Criteria:

* Unable to undergo examinations due to disturbances of consciousness or medical conditions
* Severe dementia, apraxia, disturbances of sensation or perception
* Serious complications including severe heart failure, hepatic dysfunction, renal insufficiency,or shock
* Parkinson's disease, malignant tumor, autoimmune diseases

Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Study Population: chronic-stage patients of unilateral middle cerebral artery infarction
Sampling Method: Non-Probability Sample
Enrollment: 80 (Estimated)
Dates: Start 2008-09; Primary Completion 2009-07 (Estimated)

CONTACTS AND LOCATIONS:
Overall Officials: Wei Wang, Doctor, Principal Investigator — Tongji Hospital
Locations (1):
- Department of Neurology of Tongji Hospital, Huazhong University of Science and Technology, Wuhan, Hubei, China